CLINICAL TRIAL: NCT03120715
Title: Comparison of Clinical Pregnancy Rates Between Two Protocols, With or Without Low Molecular Weight Heparin Administration Before Frozen Embryo Transfer in Hormonal Replacement Cycles: a Prospective Randomized Controlled Trial
Brief Title: Pregnancy Outcome of Women Using Low Molecular Weight Heparin Before Frozen-thawed Embryo Transfer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2017-024
Record Dates: First submitted 2017-04-05; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Infertility
Keywords: low molecular weight heparin (LMWH); frozen embryo transfer (FET); pregnancy
MeSH Terms: conditions — Infertility | interventions — Estrogens; Heparin, Low-Molecular-Weight; Chorionic Gonadotropin; Progesterone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NLMWH-A (Placebo Comparator): non-low molecular weight heparin-group A(group NLMWH-A).Without administration of low molecular weight heparin (LMWH) before FET.The oral estrogen replacement is 4mg per day (2 mg twice daily), 4 days; 6 mg per day, 4 days. Then, the patient's endometrial thickness is evaluated through vaginal ultrasound and if the endometrial thickness is <7 mm, increasing estrogen by 2 mg is given to patients until the endometrial thickness is >9 mm.If the endometrial thickness is greater than 9 mm, Human Chorionic Gonadotropin（hCG） 10000 IU will be administered via intramuscular injection.on the next day(D0), progesterone in oil 60 mg will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later(D3).
  Interventions: Drug: estrogen; Drug: hCG; Drug: progesterone
- LMWH-B (Experimental): low molecular weight heparin-group B(group LMWH-B).With administration of low molecular weight heparin (LMWH) before FET.The oral estrogen replacement is 4mg per day (2 mg twice daily), 4 days; 6 mg per day, 4 days. Then, the patient's endometrial thickness is evaluated through vaginal ultrasound and if the endometrial thickness is <7 mm, increasing estrogen by 2 mg is given to patients until the endometrial thickness is >9 mm.If the endometrial thickness is greater than 9 mm, Human Chorionic Gonadotropin（hCG） 10000 IU will be administered via intramuscular injection.on the next day(D0), progesterone in oil 60 mg will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later(D3).
  Interventions: Drug: estrogen; Drug: Low Molecular Weight Heparin; Drug: hCG; Drug: progesterone

INTERVENTIONS:
Drug: estrogen — The oral estrogen replacement is 4mg per day (2 mg twice daily), 4 days; 6 mg per day, 4 days. Then, the patient's endometrial thickness is evaluated through vaginal ultrasound and if the endometrial thickness is <7 mm, increasing estrogen by 2 mg is given to patients until the endometrial thickness is >9 mm.
  Other Names: estrodiol
Drug: Low Molecular Weight Heparin — If the endometrial thickness is greater than 9 mm, hCG 10000 IU will be administered via intramuscular injection.And low molecular weight heparin (LMWH) will be injected subcutaneously 4100 IU (WHO) every other day before FET.Then on the next day(D0), progesterone in oil 60 mg will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later(D3).
  Other Names: LMWH
  Arms: LMWH-B
Drug: hCG — If the endometrial thickness is greater than 9 mm, Human Chorionic Gonadotropin（hCG） 10000 IU will be administered via intramuscular injection.
  Other Names: Human Chorionic Gonadotropin
Drug: progesterone — on the next day(D0), progesterone in oil 60 mg will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later(D3).

SUMMARY:
Embryo freezing is a technique used commonly to optimize the pregnancy rate in assisted reproduction techniques (ART). Hormone replacement therapy (HRT) regimen is applied to prepare endometrium for frozen embryo transfer (FET) commonly.At present, It is unclear whether preimplantation low molecular weight heparin (LMWH) improves live birth and pregnancy rates in subfertile women undergoing FET. The study is a prospective randomized controlled trial to compare the pregnancy outcomes of FET in hormonal replacement therapy(HRT) cycles with or without LMWH administration before implantation.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial. Patients undergoing FET in Center for Reproductive Medicine of Nanfang Hospital, Southern Medical University are recruited.

They are randomly allocated to be prepared for transfer by using HRT cycle, with(low molecular weight heparin-group B(group LMWH-B)) or without( non-low molecular weight heparin-group A(group NLMWH-A)) administration of low molecular weight heparin (LMWH) before frozen embryo transfer (FET).

Both groups use the same protocol of HRT-FET. The oral estrogen replacement is 4mg per day (2 mg twice daily), 4 days; 6 mg per day, 4 days. Then, the patient's endometrial thickness is evaluated through vaginal ultrasound and if the endometrial thickness is <7 mm, increasing estrogen by 2 mg is given to patients until the endometrial thickness is >9 mm.In group NLMWH-A, If the endometrial thickness is greater than 9 mm, human chorionic gonadotropin (hCG)10000 IU will be administered via intramuscular injection. Then on the next day(D0), progesterone in oil 60 mg will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later(D3). In group LMWH-B, If the endometrial thickness is greater than 9 mm, hCG 10000 IU will be administered via intramuscular injection. And low molecular weight heparin (LMWH) will be injected subcutaneously 4100 IU (WHO) every other day before FET. Then on the next day(D0), progesterone in oil 60 mg will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later(D3).

This study was approved by the medicine ethics committee of Nanfang Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 to 43 years;
* Body mass index (BMI) between 19 kg/m2 and 25 kg/m2;
* At least one good quality D3 embryos for transfer;
* prepare endometrium by hormone replacement therapy(HRT)protocal;
* capable of giving informed consent.

Exclusion Criteria:

* Women or their partner with abnormal chromosome karyotype including chromosome polymorphism;
* Women diagnosed as uterus abnormality: malformed uterus (uterus unicorns, septate uterus, duplex uterus, uterus bicornis), adenomyosis, submucous myoma, intrauterine adhesion;
* Women who underwent unilateral ovariectomy or with history of ovarian tumor surgery ;
* infection factors: TORCH virus (including Toxoplasma virus, rubella virus, cytomegalovirus,herpes simplex infection),Chlamydia and Mycoplasma, etc;
* Endometriosis;
* Having hydrosalpinx ;
* Low molecular weight heparin contraindications: thrombocytopenia, hemophilia and other bleeding disorders, liver and kidney dysfunction, with a clear history of heparin allergy or allergic constitution, etc.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 342 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-09-05 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4-6 weeks
  The pregnancy rate will be evaluated in patients of each groups 4-6 weeks after embryo transfer.

SECONDARY OUTCOMES:
Implantation rate | 4-6 weeks
  Evaluation the implantation rate in patients of each groups 4-6 weeks after frozen embryo transfer
Ongoing pregnancy | 12 weeks
  Evaluation the ongoing pregnancy by monitoring pregnant bursa and fetal heart through ultrasound in patients of each group 12 weeks after embryo transfer.
miscarriage rate | Evaluation the miscarriage rate in patients of each group 12 weeks after embryo transfer.
  12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, M.D, Ph.D, Principal Investigator — Center for Reproductive Medicine, Department of Obstetrics and Gynecology, Nanfang Hospital, Southern Medical University
Locations (1):
- Center for Reproductive Medicine, Department of Obstetrics and Gynecology, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided